CLINICAL TRIAL: NCT05746585
Title: The TALK; A Novel Nurse-led, Family-based Web-based Application Marketed in Barbershops and Beauty Salons for Black Fathers and Mothers to Promote Sexual Health Among Black Male Adolescents and Young Adults in the United States
Brief Title: The TALK for Black Male Adolescent Sexual Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00105116
Record Dates: First submitted 2023-01-23; First posted 2023-02-27 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Sexuality Education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The TALK intervention for Black male adolescents and young adults (AYA) (Experimental): The TALK, a parent-centered, adolescent-involved health promotion intervention for Black male adolescents and young adults (AYA). Through the use of entertainment videos and educational modules, investigators will provide parents with resources and tools for communicating with their adolescents about sexual health and experiences of racial discrimination, and how these experiences impact sexual health.
  Interventions: Behavioral: The Talk Web-based resources

INTERVENTIONS:
Behavioral: The Talk Web-based resources — Educational videos and podcasts for parents and their sons

SUMMARY:
The purpose of this study is to construct the first nurse-led web-based intervention, The TALK, a parent-centered, adolescent-involved health promotion intervention for Black male adolescents and young adults (AYA). Through the use of entertainment videos and educational modules, investigators will provide parents with resources and tools for communicating with their adolescents about sexual health and experiences of racial discrimination, and how these experiences impact sexual health.

ELIGIBILITY:
Inclusion Criteria:

Self-identified as a parent, parent figure, or caregiver of a Black or African American male adolescent between the ages of 13-17 years, able to speak and read English. Adolescents of these parents will also be recruited along with their parents. Adolescents recruited will be required to sign additional consent forms.

Exclusion Criteria:

-

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Usability | 6 months
  Usability of The TALK as measured by number of website uses
Acceptability | 6 months
  Acceptability of The TALK as measured by participant survey feedback
Communication Frequency | 6 months
  Frequency of parent-adolescent sexual health communication measured by survey feedback
Communication Quality | 6 months
  Quality of parent-adolescent sexual health communication as measured by survey feedback

CONTACTS AND LOCATIONS:
Overall Officials: Schenita Randolph, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No